CLINICAL TRIAL: NCT06162598
Title: The Effect of Preparation With The Ventriloquist Puppet Method Before Inhaler Treatment on Anxiety and Fear Level of Children Aged 4-6
Brief Title: The Ventriloquist Puppet Method for Children Under The Inhaler Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Tuba Arpacı, Asisstant Professor, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KMU-SBF-TA-02
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-11

CONDITIONS: Hospitalism in Children
Keywords: Children; Nursing; Puppet; Ventriloquist; Inhaler treatment; Therapeutic approach

STUDY DESIGN:
Intervention Model Description: Two group with conventional therapy control group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Children in the control group will undergo the routine preparation procedure applied in the emergency department. Before and after inhaler treatment, the child, parent, and nurse will be asked to fill out data collection forms to assess the child's anxiety and fear levels.
- Ventriloquist Puppet group (Experimental): The preparation for the procedure will be accompanied by a puppet before the treatment. The child will be told about the features of the puppet and will be introduced to it. The inhaler treatment application will be explained to the intervention group through the ventriloquist puppet method. By making the puppet talk using the ventriloquism technique, the child will be able to understand the procedure. The application of the inhaler will be shown to the child with the help of a nebulizer mask on the puppet. Before the application and after the inhaler treatment, the child, parent, and nurse will be asked to fill out the children's state anxiety scale and children's fear scale to evaluate the child's anxiety and fear levels.
  Interventions: Other: Ventriloquist Puppet

INTERVENTIONS:
Other: Ventriloquist Puppet — one day preparation intervention applied by researcher for children under the inhaler treatment. Preparation will be 30 minutes long
  Arms: Ventriloquist Puppet group

SUMMARY:
This study aimed to determine the effect of preparation with the ventriloquist puppet method before inhaler treatment on anxiety and fear level of children aged 4-6

DETAILED DESCRIPTION:
Although treatment methods appropriate to the disease are applied in respiratory system diseases, healthcare professionals must cooperate with the child and family regarding compliance with the treatment (oral, nebulizer, inhaler) and management of the disease. Children may experience anxiety and fear from the moment they enter the hospital. They may react to being in the hospital and medical procedures such as crying, running away, or withdrawing. Age, previous negative hospitalization experiences, and fear of getting sick are factors that shape children's medical fears. The majority of children have 'a little' or 'a lot' of fear about medical procedures. Children have adaptation problems to the inhaler treatment and often reject it. To provide effective treatment, compliance of the child and family with the treatment and suitable application techniques are crucial. In this process, it is important to minimize the anxiety and fear of children and ensure that they receive the treatment in the best possible way. Therapeutic approaches such as distraction cards, musical toys, and puppets during the preparation of the child for the procedure before the treatment can increase the child's compliance with the treatment and reduce the level of anxiety. In a study, puppet shows were useful in reducing the fears of children with 'a lot' fear. In another study, finger puppets as a play enhanced communication with children with cancer and were suitable for use in the hospital environment. It has been concluded that the use of puppets is beneficial because it gives children the opportunity to express themselves freely. An effort should be made to reduce the child's anxiety and fear by taking a therapeutic approach not only for invasive procedures but also for non-invasive procedures. Therapeutic approaches can be applied to the child and family before, during, and after treatment. This study aimed to determine the effect of preparation with the ventriloquist puppet method before inhaler treatment on the anxiety and fear levels of children aged 4-6.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4-6,
* Children receiving inhaler therapy,
* Children and families who can speak Turkish,
* Children and families who volunteer to participate in the research,

Exclusion Criteria:

* Children with cognitive or mental problems,
* Children with life-threatening conditions,
* Children with hearing, vision and/or speech impairments

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety | one day
  Children's State Anxiety Scale: Validated scale used for evaluation of 4-10 aged children's anxiety level. Scale score ranges between 0-10
Fear | one day
  Children's Fear Scale: Validated scale used for evaluation of 5-10 aged children's fear level. Scale score ranges between 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba ARPACI, PhD, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Tuba ARPACI, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No